CLINICAL TRIAL: NCT02250105
Title: Trial of ARI-3037MO to Reduce Triglyceride Levels in Adults With Severe (≥500 mg/dl) Hypertriglyceridemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arisaph Pharmaceuticals Inc (Industry)
Collaborators: Baim Institute for Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARI-3037MO-004
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2015-08

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARI-3037MO (Active Comparator): ARI-3037MO 3g bid orally for 12 weeks
  Interventions: Drug: ARI-3037MO
- Placebo (Placebo Comparator): Matching placebo 3g bid orally for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARI-3037MO — Lipid lowering
  Arms: ARI-3037MO
Drug: Placebo — Inactive
  Arms: Placebo

SUMMARY:
This study is to evaluate the efficacy and safety of ARI-3037MO 3g BID compared to placebo in reducing triglyceride (TG) levels of subjects with severe (≥500 mg/dL and <2,000 mg/dL) hypertriglyceridemia. Eligible patients will enter a 4- to 6-week lead-in period (6-week washout for subjects on non-statin lipid-lowering therapy [subjects may remain on statins during this period], 4 weeks for patients on statins only or not receiving any type of lipid-lowering therapy), followed by qualifying fasting TG measurements at visits 2 and 3, at least 7 days apart. If the baseline TG value is > 500 mg/dL and < 2,000 mg/dL, the qualified subjects will be randomized at visit 4 and enter the double-blind, 12-week efficacy and safety assessment phase. End-of-study lipid levels will be assessed on visits 6 and 7 (weeks 11 and 12 average). A final closeout and safety assessment visit will be done 14 weeks post randomization

ELIGIBILITY:
Inclusion Criteria 1. Age ≥ 18 years. 2. Subjects willing to comply with lifestyle intervention modifications (diet and exercise) 3. TG levels: At randomization, mean level > 500 mg/dL and < 2,000 mg/dL. 4. Understands the trial requirements and the treatment procedures, is willing to comply with all protocol-required follow-up evaluation and provides written informed consent.

5. Patients already taking statin therapy must be on a stable dose, defined as no changes in the dose of statin in the 3 months prior to enrollment, and must be willing and able to remain on that dose for the duration of the study.

-

Exclusion Criteria 1. History of pancreatitis. 2. Body mass index > 45 kg/m2. 3. Weight change ≥ 3 kg during the lead-in period. 4. Contraindication to niacin treatment (prior flushing is not regarded as a contraindication to niacin treatment).

5. Uncontrolled diabetes, defined as HbA1C > 10.5. 6. Subjects who would benefit from statin treatment per clinical guidelines but who are not taking statins are excluded. However, these patients may be included only if the subject's primary care physician confirms the decision not to treat according to guidelines and its reason (e.g. statin intolerant subjects, subject refusal, etc.), and it has been agreed upon by the subject, the site investigator, and the primary care physician, after discussion of the potential risks of non-treatment with statins..

7. History of stroke, myocardial infarction, life-threatening arrhythmia, or coronary vascularization within 6 months before screening.

8. Thyroid-stimulating hormone ≥ 1.5 times the ULN. 9. Clinical evidence of hypothyroidism or thyroid hormonal therapy that has not been stable for ≥ 6 weeks before screening.

10. Creatine kinase concentration ≥ 3 times the ULN. 11. Known, active liver disease, including but not limited to:

1. Confirmed alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, or bilirubin ≥ 2 times the ULN.
2. Hepatitis C (anti-hepatitis C virus IgG +).
3. Hepatitis B (hepatitis B surface [HBs] antigen +, anti hepatitis B core [HBc] antigen immunoglobulin M [IgM]+).
4. Hepatitis A (anti HBa IgM+). 12. Blood donation of ≥ 1 pint (0.5 L) within 30 days before screening or plasma donation within 7 days before screening.

   13. History of symptomatic gallstone disease unless treated with cholecystectomy.

   14. Known nephrotic syndrome or ≥ 3 g/day proteinuria. 15. Past organ transplant or on a waiting list for an organ transplant. 16. Currently receiving or scheduled to receive chemotherapy within 30 days before or after enrollment.

   17. Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 12 months.

   18. Problems with substance abuse, which, in the opinion of the investigator, might affect study compliance.

   19. Planned procedure that may cause non-compliance with the protocol or confound data interpretation.

   20. Current participation in another investigational drug or device clinical trial that has not reached its primary endpoint.

   21. Women who intend to become pregnant within 12 months after enrollment. Women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after enrollment.

   22. Women who are pregnant or nursing. 23. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Triglyceride levels | 12 weeks

SECONDARY OUTCOMES:
Change in LDL cholesterol | 12 weeks
Change in HDL cholesterol | 12 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Orange County Research Center, Tustin, California
  - Louisville Metabolic and Atherosclerosis Research Center, Louisville, Kentucky
  - Maine Research Associates, Auburn, Maine
  - Sterling Clinical Research Inc, Cincinnati, Ohio
  - National Clinical Research inc, Richmond, Virginia